CLINICAL TRIAL: NCT03530566
Title: Prospective Comparative Clinical Study to Evaluate Effectiveness of a Standardized Multidisciplinary Weight Loss Program in Obese Patients During 3 Months Prior to Bariatric Surgery
Brief Title: Study to Evaluate Effectiveness of a Weight Loss Program in Obese Patients During 3 Months Prior to Bariatric Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Protein Supplies SL (Other)
Responsible Party: Sponsor
Other Study IDs: PRO-CBP-2017-02
Record Dates: First submitted 2018-05-08; First posted 2018-05-21 (Actual); Last update posted 2018-05-24 (Actual); Status verified 2018-05

CONDITIONS: Obesity, Morbid; Bariatric Surgery; Comorbidity
Keywords: PnK Method; obesity; very low calorie ketogenic diet; Comorbidity; Bariatric Surgery; weight loss
MeSH Terms: conditions — Obesity, Morbid; Obesity; Weight Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pnk group: Patients with morbid obesity (BMI ≥ 40 kg/m2) or with severe obesity (BMI 35 to 39.9 kg/m2), with two or more comorbidities, scheduled bariatric surgery within 3 months will be treated with PnK® Method
  Interventions: Other: PnK® Method
- Control group: Patients with morbid obesity (BMI ≥ 40 kg/m2) or with severe obesity (BMI 35 to 39.9 kg/m2), with two or more comorbidities, treated with standard diet 3 moths prior bariatric surgery
  Interventions: Other: standard diet

INTERVENTIONS:
Other: PnK® Method — A multidisciplinary program of weight loss based on diet (initially very low ketogenic diet), physical activity and emotional support
  Groups: Pnk group
Other: standard diet — standard low calorie diet for weight loss
  Groups: Control group

SUMMARY:
Prospective multicenter observational clinical study on a dietary regimen in obese patients scheduled for bariatric surgery.

DETAILED DESCRIPTION:
Study population: 25 patients with morbid obesity (BMI ≥ 40 kg / m2) or severe obesity (BMI 35 to 39.9 kg / m2) , with two or more comorbidities, scheduled for bariatric surgery within 3 months, and who will start treatment with the multidisciplinary weight loss program (PnK Method) based on diet, exercise and psychological support.

Patients will be followed-up for 3 months, with the following controls: pre-selection, baseline, month 1, month 2, month 3, and control when hospital discharge.

The treatment schedule in these patients will be as follows: a very low calorie ketogenic diet for at least 1 month or until losing 10% of the weight, and then, a low calorie diet with gradual reintroduction of natural foods for 2 months, until surgery.

The investigators will obtain retrospective data from 25 patients treated with the standard diet who met the same inclusion/exclusion criteria as the patients in this study and who similarly resemble in age, sex and BMI, for comparative analysis (control group).

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes, between 18 and 65 years old
* Patients with morbid obesity (BMI ≥ 40 kg/m2) or with severe obesity (BMI 35 to 39.9 kg/m2), with two or more comorbidities associated with obesity (type 2 diabetes mellitus, arterial hypertension, obstructive sleep apnea, obesity hypoventilation syndrome, chronic respiratory disease, metabolic syndrome, atrial fibrillation, heart failure, pulmonary hypertension, cardiomyopathy, history of thrombosis, renal failure).
* Patients scheduled for bariatric surgery within 3 months ± 1 week.
* Patients who, regardless of their inclusion in this study, will undergo treatment with the multidisciplinary slimming program in study or standard diet.
* Patients who agree to participate and sign the Informed Consent

Exclusion Criteria:

* Pregnant or lactating women.
* Patients with type 1 diabetes mellitus or on insulin therapy
* Patients with eating disorders, alcoholism, and/or drug addiction.
* Patients with any severe psychological disorder (eg schizophrenia, bipolar disorder).
* Patients receiving dicumarinic anticoagulants (Sintrom®) or cortisone.
* Patients with liver failure.
* Patients with severe kidney failure (gfr <30).
* Patients with hemopathies.
* Patients with cancer.
* Patients with cardiovascular or cerebrovascular disease (heart rate disorders, recent infarction [<6m], unstable angina, decompensated heart failure, recent stroke [<6m]).
* Patients in acute attack of gout.
* Patients with renal lithiasis verified by ultrasound.
* Patients with cholelithiasis verified by ultrasound.
* Patients with depression.
* Patients with electrolyte imbalance, according to medical criteria.
* Patients with orthostatic hypotension.
* Patients with contraindications to surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with morbid obesity (BMI ≥ 40 kg/m2) or with severe obesity (BMI 35 to 39.9 kg/m2), with two or more comorbidities, scheduled to undergo bariatric surgery within 3 months, should be treated with the multidisciplinary weight loss program in study.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2018-05 (Estimated); Primary Completion 2019-01 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Body weight loss at 3 monthes | from baseline to 3 monthes
  Change in body weight from baseline to 3 monthes

SECONDARY OUTCOMES:
Body weight loss at 2 monthes | from baseline to 2 monthes
  Change in body weight from baseline to 2 monthes
Body weight loss at 1 month | from baseline to 1 month
  Change in body weight from baseline to 1 month
Change in systolic blood pressure at 3 monthes | from baseline to 3 monthes
  Change in systolic blood pressure from baseline to 3 monthes
Change in diastolic blood pressure at 3 monthes | from baseline to 3 monthes
  Change in diastolic blood pressure from baseline to 3 monthes
Change in systolic blood pressure at 2 monthes | from baseline to 2 monthes
  Change in systolic blood pressure from baseline to 2 monthes
Change in diastolyc blood pressure at 2 monthes | from baseline to 2 monthes
  Change in diastolyc blood pressure from baseline to 2 monthes
Change in systolic blood pressure at 1 month | from baseline to 1 month
  Change in systolic blood pressure from baseline to 1 month
Change in diastolic blood pressure at 1 month | from baseline to 1 month
  Change in diastolic blood pressure from baseline to 1 month
Change in blood glucose at 3 monthes | from baseline to 3 monthes
  Change in blood glucose level from baseline to 3 monthes
Change in blood glucose at 2 monthes | from baseline to 2 monthes
  Change in blood glucose level from baseline to 2 monthes
Change in blood glucose at 1 month | from baseline to 1 month
  Change in blood glucose level from baseline to 1 month
Change in HbA1c at 3 monthes | from baseline to 3 monthes
  Change in HbA1c (Glycated hemoglobin) percentage from baseline to 3 monthes
Change in HbA1c at 2 monthes | from baseline to 2 monthes
  Change in HbA1c (Glycated hemoglobin) percentage from baseline to 2 monthes
Change in HbA1c at 1 month | from baseline to 1 month
  Change in HbA1c (Glycated hemoglobin) percentage from baseline to 1 month
Change in total cholesterol level at 3 monthes | from baseline to 3 monthes
  Change in blood total cholesterol level from baseline to 3 monthes
Change in total cholesterol level at 2 monthes | from baseline to 2 monthes
  Change in blood total cholesterol level from baseline to 2 monthes
Change in total cholesterol level at 1 month | from baseline to 1 month
  Change in blood total cholesterol level from baseline to 1 months
Change in triglycerides level at 3 monthes | from baseline to 3 monthes
  Change in blood triglycerides level from baseline to 3 monthes
Change in triglycerides level at 2 monthes | from baseline to 2 monthes
  Change in blood triglycerides level from baseline to 2 monthes
Change in triglycerides level at 1 month | from baseline to 1 month
  Change in blood triglycerides level from baseline to 1 month
Metabolic Control of type 2 Diabetes at 3 months | from baseline to 3 monthes
  Percentage of patients with better, equal or worse metabolic control of type 2 Diabetes at 3 months regarding baseline
Clinical Control of arterial hypertension at 3 months | from baseline to 3 monthes
  Percentage of patients with better, equal or worse clinical control of arterial hypertension at 3 months regarding baseline
Clinical Control of Hypercholesterolemia at 3 months | from baseline to 3 monthes
  Percentage of patients with better, equal or worse clinical control of Hypercholesterolemia at 3 months regarding baseline
Clinical Control of Hypertriglyceridemia at 3 months | from baseline to 3 monthes
  Percentage of patients with better, equal or worse clinical control of Hypertriglyceridemia at 3 months regarding baseline
Improvement of Sleep Apnea Obstructive Syndrome at 3 months | from baseline to 3 monthes
  Percentage of patients with better, equal or worse clinical symptoms of Sleep Apnea Obstructive Syndrome, regarding baseline.
Improvement of Chronic Respiratory Disease at 3 months | from baseline to 3 monthes
  Percentage of patients with better, equal or worse clinical symptoms of Chronic Respiratory Disease, regarding baseline.
Improvement of Obesity hypoventilation syndrome at 3 months | from baseline to 3 monthes
  Percentage of patients with better, equal or worse clinical symptoms of Obesity hypoventilation syndrome, regarding baseline.
Improvement of Metabolic syndrome at 3 months | from baseline to 3 monthes
  Percentage of patients with better, equal or worse clinical symptoms of Percentage of patients with better, equal or worse clinical symptoms of Obesity hypoventilation syndrome, regarding baseline.
Improvement of Atrial fibrillation at 3 months | from baseline to 3 monthes
  Percentage of patients with better, equal or worse clinical symptoms of Atrial fibrillation, regarding baseline.
Improvement of Cardiac insufficiency at 3 months | from baseline to 3 monthes
  Percentage of patients with better, equal or worse clinical symptoms of Cardiac insufficiency, regarding baseline.
Improvement of Pulmonary hypertension at 3 months | from baseline to 3 monthes
  Percentage of patients with better, equal or worse clinical symptoms of Pulmonary hypertension, regarding baseline.
Improvement of Cardiomyopathy at 3 months | from baseline to 3 monthes
  Percentage of patients with better, equal or worse clinical symptoms of cardiomyopathy, regarding baseline.
Improvement of Renal insufficiency at 3 months | from baseline to 3 monthes
  Percentage of patients with better, equal or worse clinical symptoms of Renal insufficiency, regarding baseline.
Obesity Surgery Mortality Risk Score | 3 months
  Obesity Surgery Mortality Risk Score at the preoperative visit
Length of surgery | During bariatric surgery
  Length (in minuts) of bariatric surgery
Length of anesthesia | During bariatric surgery
  Length (in minuts) of anesthesia during bariatric surgery
Number of patients with intraoperative complications | During bariatric surgery
  Number of patients with intraoperative complications occurring during bariatric surgery and within the postoperative 24 hours
Number of patients with postoperative complications after bariatric surgery | After bariatric surgery
  Number of patients with postoperative complications occurring before hospital discharge
Number of total days of hospitalization | After bariatric surgery
  Number of total days of hospitalization after bariatric surgery
Number of Participants With Adverse Events related to preoperative weight loss treatment | Through 3 months of study
  Number of Participants with Adverse Events as a Measure of Safety and Tolerability of standardized weight-loss programme (PnK® Method)
Number of weight loss treatment dropout rate | from baseline to 3 monthes
  Number of weight loss treatment dropout rate from baseline to 3 months
Number of patients who refuse bariatric surgery at 3 months | from baseline to 3 monthes
  Number of patients who refuse bariatric surgery from baseline to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Davide De Carvalho, Ph, Principal Investigator — Centro Hospitalar Sao Joao do Porto; Paula Freitas, Ph, Principal Investigator — Centro Hospitalar Sao Joao do Porto